CLINICAL TRIAL: NCT03057561
Title: Efficacy of Dotarem® (Gd-DOTA) Versus Gadovist® (Gd-DO3A-butrol) for Late Gadolinium Enhancement Cardiac Magnetic Resonance and Relationship to Outcomes: A Pilot Study
Brief Title: Efficacy of Dotarem® (Gd-DOTA) Versus Gadovist® (Gd-DO3A-butrol) for Late Gadolinium Enhancement Cardiac Magnetic Resonance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Dipan Shah (Other)
Collaborators: Guerbet (Industry)
Responsible Party: Sponsor-Investigator, Dipan Shah, Director, Cardiac Magnetic Resonance Imaging, The Methodist Hospital Research Institute
Organization: The Methodist Hospital Research Institute (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: Pro00012234
Record Dates: First submitted 2017-01-18; First posted 2017-02-20 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Coronary Artery Disease; Cardiomyopathy
Keywords: CAD
MeSH Terms: conditions — Coronary Artery Disease; Cardiomyopathies | interventions — gadoterate meglumine; gadolinium 1,4,7,10-tetraazacyclododecane-N,N',N'',N'''-tetraacetate; Contrast Media; Product Labeling; gadobutrol

STUDY DESIGN:
Intervention Model Description: Evaluating the efficacy of Dotarem enhanced MRI compared to Gadovist enhanced MRI in identifying myocardial fibrosis. Patients will be randomized (in a 1:1 fashion) to receive either Dotarem or Gadovist for LGE-CMR such that there will be 60 patients in the Dotarem cohort and 60 patients in the Gadovist cohort
Who Masked: Outcomes Assessor
Masking Description: Blinded reader of scans will not know whether subject received Dotarem or Gadovist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3.0 Tesla Cardiac MRI using Dotarem contrast agent (Experimental): 60 randomly selected participants with suspected or known cardiovascular disease will have a 3.0 Tesla Cardiac MRI with contrast agent, Dotarem
  Interventions: Drug: Cardiac MRI taken using contrast agent, Dotarem® (Gd-DOTA); Drug: Cardiac MRI with contrast agent, Gadovist
- 3.0 Tesla Cardiac MRI using a Gadovist contrast agent (Experimental): 60 randomly selected participants with suspected or known cardiovascular disease will have a 3.0 Tesla Cardiac MRI with contrast agent, Gadovist
  Interventions: Drug: Cardiac MRI taken using contrast agent, Dotarem® (Gd-DOTA); Drug: Cardiac MRI with contrast agent, Gadovist

INTERVENTIONS:
Drug: Cardiac MRI taken using contrast agent, Dotarem® (Gd-DOTA) — Gadolinium based contrast agent used in cardiac MRI scanning using 3.0 Tesla MRI
  Other Names: Cardiac MRI with contrast; CMR with tracer or contrast agent; Dotarem (Gd-DOTA) contrast agent
Drug: Cardiac MRI with contrast agent, Gadovist — Brand of Gd-DO3A-butrol; contrast agent used in cardiac MRI scanning using 3.0 Tesla MRI
  Other Names: Cardiac MRI with contrast; CMR with tracer or contrast agent; Gadovist® (Gd-DO3A-butrol) contast agent

SUMMARY:
This project is designed to demonstrate equivalence of Dotarem enhanced LGE-CMR (late gadolinium enhancement cardiac MRI) with Gadoviost enhanced LGE-CMR from the standpoint of visual image quality, quantitative image quality, and association with clinical outcomes.

DETAILED DESCRIPTION:
Gadolinium-containing contrast agents (GdCAs) are intravenous agents used for contrast enhancement with magnetic resonance imaging (MRI) and with magnetic resonance angiography (MRA). The GdCAs (gadodiamide, gadopentetic acid, gadobenic acid, gadoxetic acid, gadoteridol, gadobutrol and gadoteric acid) have been in use for few decades for different types of MR scan varying from product to product, including liver, brain, and whole body scan.

Recently, there has been a great interest in employing contrast-related techniques to assess for fibrosis in the myocardium of the heart. As opposed to nuclear methods, viability assessment by MRI is a nonstress examination that provides high-resolution detail, including functional assessment of the left ventricle in approximately 30 minutes. Assessment of myocardial viability is performed using 5- to 20-minute delayed, gadolinium-enhanced MRI. On delayed MRI, there is a relatively decreased washout of the gadolinium contrast agent in areas of myocardium that have been replaced by fibrosis or scar. In normal viable myocardium, the gadolinium contrast agent washes out more rapidly than it does from the fibrosis or scar. Since the difference between normal and abnormal myocardium is based on washout kinetics, images that are delayed by 5 to 20 minutes after contrast injection will optimally depict the fibrosis or scar.

The differences in gadolinium enhancement on MRI of viable myocardium and fibrosis or scar have been known for many years. Recently, however, MRI pulse sequences have been developed that greatly improve the conspicuity of the enhanced areas of myocardium that have been replaced by fibrosis or scar. The pulse sequence used is an inversion-recovery prepared gradient-echo sequence. In this method, an inversion pulse is used to null the signal from normal myocardium. Myocardium that is replaced by fibrosis or scar retains gadolinium and shows very high signal intensity compared with the suppressed, darker myocardium.

Gadovist has been the standard gadolinium contrasts used in the U.S. in CMR imaging for the past few years. On the other hand, Dotarem, a widely used contrast agent in Europe, has been introduced to be used in the U.S. market.The sensitivity of Dotarem to that of Magnevist in determining the location and extent of scar in patients scanned with CMR will be Gadovist in this study.

The CMR laboratory at the Houston Methodist DeBakey Heart & Vascular Center is one of the largest dedicated CMR laboratories in the U.S. performing 3,000 clinical CMR procedures per year. The laboratory has been in existence since 2008 and is currently equipped with 2 dedicated MRI scanners: 1.5T Siemens Avanto and 3.0T Siemens Verio. Through a research agreement with Siemens Medical Solutions, the laboratory has access to numerous works-in progress sequences as they are developed. The laboratory is equipped with an MRI compatible patient monitoring system, infusion pump, and power injector and is staffed by a team of 5 dedicated CMR technologists, 2 clinical nurses, 1 CMR fellow, an MRI scientist, and 2 attending cardiologists.

One hundred twenty patients with known or suspected cardiovascular disease will be recruited for this study. Patients will be randomized (in a 1:1 fashion) to receive either Dotarem or Gadovist for LGE-CMR such that there will be 60 patients in the Dotarem cohort and 60 patients in the Gadovist cohort.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing clinically referred CMR.

Exclusion Criteria:

1. Patients who are unable to give informed consent.
2. Individuals with severe claustrophobia.
3. Individuals unable to lie flat for 90 minutes (the anticipated amount of time to complete the MRI procedure).
4. Individuals who are pregnant.
5. Patients with implants or pacemakers.
6. Patients that have hypersensitivity to components of gadolinium.
7. Patients with renal failure.
8. Patients who had any trauma or surgery which may have left ferromagnetic material in the body.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-10-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Compare visual image quality of LGE-CMR when performed with Dotarem or Gadovist in a randomized fashion. | Two years
  All LGE-CMR scans scoring for visual image quality using a 5-point scale: 1 = LV myocardium not visible, 2 = severe artifact interfering with ability to visualize LV myocardial borders limiting assessment for presence of LGE (poor), 3 = LV myocardial borders are well delineated but there is moderate artifact affecting ability to identify LGE (fair), 4 = LV myocardium is well delineated with minor artifacts affecting ability to identify LGE (good), 5 = LV myocardium well delineated with no artifacts affecting ability to identify LGE (excellent).
Compare quantitative signal enhancement of LGE when performed with Dotarem or Gadovist in a randomized fashion. | Two Years
  Assessment of the intensity of hyperenhancement with Dotarem and Gadovist using a semi-automated computer software.
Compare association of LGE and clinical cardiovascular outcomes when performed with Dotarem or Gadovistin a randomized fashion. | Eight years
  Patient screened for outcomes (e.g. acute myocardial infraction, sudden cardiac death, heart failure, stroke, cardiovascular hemorrhage, other death from cardiovascular causes)

CONTACTS AND LOCATIONS:
Overall Officials: Dipan Shah, MD, Principal Investigator — The Methodist Hospital Research Institute

IPD SHARING:
Plan to Share IPD: Undecided